CLINICAL TRIAL: NCT02132247
Title: An Open-label, Prospective, Uncontrolled Study of the Safety and Local Tolerability of the Diclofenac Epolamine Patch (Flector Patch) in Pediatric Patients With Minor Soft Tissue Injuries
Brief Title: Safety Study of Flector Patch in Children With Minor Soft Tissue Injuries
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: IBSA Institut Biochimique SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08US/Fp03
Record Dates: First submitted 2014-04-28; First posted 2014-05-07 (Estimated); Results first posted 2018-05-11 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-04

CONDITIONS: Athletic Injuries
Keywords: Minor athletic injuries; Pain; Diclofenac; Topical
MeSH Terms: conditions — Athletic Injuries; Pain | interventions — diclofenac hydroxyethylpyrrolidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Flector Patch (Experimental): Flector Patch is a transdermal delivery system containing 180 mg of diclofenac hydroxyethylpyrrolidine. The patch will be used twice-a-day for up to two weeks, or until pain resolution, whichever comes first.
  Interventions: Drug: Diclofenac hydroxyethylpyrrolidine

INTERVENTIONS:
Drug: Diclofenac hydroxyethylpyrrolidine
  Other Names: Flector Patch

SUMMARY:
The primary purpose of this study is to determine whether Flector Patch is safe for use in children. The secondary purpose is to assess blood levels of diclofenac, the active ingredient in Flector Patch.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 to 16 years, either gender
* Informed consent: 6-9 year olds must have their parent/legally authorized representative complete a Parental Permission Form; 10-16 year olds must complete a Children's Assent Form and have their parent/legally authorized representative complete a Parental Permission Form
* Minor soft tissue injury within 96 hours of study entry
* Spontaneous pain of at least moderate intensity (i.e. pain of at least 3 on the 6-point Wong- Baker Faces scale for pain severity assessment by patient)
* Injury must be considered by the Investigator to be clinically significant
* Negative urine pregnancy test at screening for female subjects of childbearing potential (started the menstrual cycle)
* Able to read and speak English
* Available with their parents for the immediate two week period following study enrollment

Exclusion Criteria:

* Major soft tissue injury (Fractures are only exclusionary if the injury is stabilized with a device, e.g. a hard cast, that cannot be removed to allow a patch to be applied to the site of injury)
* Open skin lesion or any dermatological condition (e.g. skin infection, eczema) within the injured area
* Injury is midline or involves the spine, digits or hands
* Prior injury to the same site within the past 3 months
* Three or more other prior injuries (minor or major) to the region in the past
* Injury occurred more than 96 hours prior to study entry
* Prior use of topical medication to involved area within 48 hours of study entry
* Allergic disorders, including asthma or urticaria, but only if associated with exposure to aspirin or an NSAID
* Coagulation defects
* Prior use of over-the-counter (OTC) analgesics or short-acting non-steroidal anti-inflammatory drugs (NSAIDs [ibuprofen, ketoprofen]) within 6 hours of study entry (acetaminophen permitted up until the time of study entry)
* Prior use of narcotic analgesics within 7 days of study entry
* Prior use of systemic anti-inflammatory steroidal drugs within 60 days of study entry
* Prior use of long-acting NSAIDs such as piroxicam or naproxen since injury
* Concomitant use of drugs which may be susceptible to interactions with diclofenac, or affect safety if used concomitantly (serotonin-selective reuptake inhibitors (SSRI), lithium, digoxin, anticoagulants, antidiabetic agents, cyclosporin, methotrexate, quinolone antimicrobials, other NSAIDs, steroids and diuretics)
* Subjects suffering from psychiatric disorders (including depression)
* Handicapped patients, but only if the handicap prevents them from either assessing their pain or safely using the patch (e.g., pervasive developmental disorders such as autism, Asperger syndrome, Rett syndrome, Heller's syndrome, severe attention deficit hyperactivity disorders (ADHD), other severe mental retardation of traumatic, congenital or other origin)
* History of current alcohol or drug abuse dated < 1 year
* Severe cardiac, renal or hepatic impairment
* Severe systemic diseases (e.g. cancer, severe acute infection)
* Any underlying disease or medication that severely compromise the patient's immune system
* Prior history of any chronic pain disorder
* Prior history of GI bleeds/ulcers, liver or kidney disease
* Hypersensitivity to diclofenac or other NSAID drugs (including aspirin)
* Females who are pregnant or breast feeding
* Patients participating or having been involved in other clinical investigations during the three months preceding the entry of this study

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 104 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clarence Jones, Ph.D., Study Director — IBSA Institut Biochimique SA
Locations (10):
- United States (10):
  - Applied Research Center of Arkansas, Little Rock, Arkansas
  - SCORE Physician Alliance, St. Petersburg, Florida
  - Pediatrics and Adolescent Medicine P.A., Marietta, Georgia
  - Arlington Family Research Center Inc., Arlington, Texas
  - Utah Valley Pediatrics, Orem, Utah
  - J. Lewis Research Inc./Foothill Family Clininc, Salt Lake City, Utah
  - J. Lewis Research Inc./FirstMed East, Salt Lake City, Utah
  - J. Lewis Research Inc./Foothill Family Clinic South, Salt Lake City, Utah
  - Legacy Point Family Medicine, West Point, Utah
  - Pediatric Research of Charlottesville, Charlottesville, Virginia

REFERENCES:
- [Derived] Jones CA, Hoehler FK, Frangione V, Ledesma G, Wisman PP Jr, Jones C. Safety and Efficacy of the FLECTOR (Diclofenac Epolamine) Topical System in Children with Minor Soft Tissue Injuries: A Phase IV Non-randomized Clinical Trial. Clin Drug Investig. 2022 Jan;42(1):43-51. doi: 10.1007/s40261-021-01101-x. Epub 2021 Nov 26. PMID 34826122

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were no significant events in the study between enrollment (i.e. determination of eligibility) and assignment to the Flector Patch arm.
Groups:
- Flector Patch/Age 6-11; Flector Patch/Age 12-16: Flector Patch is a topical delivery system containing 180 mg of diclofenac epolamine. The patch will be used twice-a-day for up to two weeks, or until pain resolution, whichever comes first.
Period: Overall Study
Arm/Group | Flector Patch/Age 6-11 | Flector Patch/Age 12-16
Started | 52 | 52
Completed | 51 | 52
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Flector Patch/Age 6-11: 6-11 year old participants treated with Flector Patch twice per day.
- Flector Patch/Age 12-16: 12-16 year old participants treated with Flector Patch twice per day.
- Total: Total of all reporting groups
Arm/Group | Flector Patch/Age 6-11 | Flector Patch/Age 12-16 | Total
Number analyzed (Participants) | 52 | 52 | 104
Age, Customized [Count of Participants; unit: Participants] — Eligible patients between 6 and 16 years old were enrolled in equal numbers into two subgroups, 6-11 years old and 12-16 years old.
  Participants | 52 | 52 | 104
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 22 | 36
  Male | 38 | 30 | 68
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 3 | 4 | 7
  White | 42 | 43 | 85
  More than one race | 7 | 2 | 9
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 52 | 52 | 104
Injury-Associated Pain Assessment [Mean (Standard Deviation); unit: units on a scale] — Wong-Baker FACES Scale: No Hurt - 0; Hurts little bit - 1; Hurts little more - 2; Hurts even more - 3; Hurts whole lot - 4; Hurts worst - 5
  units on a scale | 3.37 (.56) | 3.58 (0.64) | 3.47 (0.61)
Height [Mean (Standard Deviation); unit: Inches] | 54.1 (4.8) | 66.4 (3.5) | 60.2 (7.4)
Weight [Mean (Standard Deviation); unit: Pounds] | 80.3 (28.1) | 149.0 (43.6) | 114.7 (50.2)

OUTCOME MEASURES:

1. Primary Outcome: Dermatologic Assessment at the Patch Application Site
Description: None - 0; Faint redness - 1; Moderate redness - 2; Intense redness - 3; Redness with edema or papules - 4; Redness with weeping vesicles, blisters or bullae - 5; Redness with extension of effect beyond margin of contact site - 6.
Time Frame: Up to 2 weeks, depending upon pain resolution
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Flector Patch/Age 6-11 | Flector Patch/Age 12-16
Number analyzed (Participants) | 52 | 52
Units on a scale
  Day1-2 | 0.10 (0.30) | 0.04 (0.19)
  Day 3-4 | 0.04 (0.20) | 0.06 (0.24)
  Day 5-7 | 0.11 (0.32) | 0.00 (0.00)
  Day 8-11 | 0.00 (0.00) | 0.06 (0.24)
  Day 12-15 | 0.00 (0.00) | 0.00 (0.00)

2. Secondary Outcome: Investigator Assessment of the Global Response to Therapy on a 5-point Scale
Description: 5-point scale: No clinical improvement in pain intensity and/or functional performance - 1; Slight clinical improvement in pain intensity and/or functional performance - 2; Moderate clinical improvement in pain intensity and/or functional performance - 3; Marked clinical improvement in pain intensity and/or functional performance - 4; Restoration of normal functional performance in the absence of any pain - 5.
Time Frame: Up to 2 weeks, depending upon pain resolution
Measure: Count of Participants; unit: Participants
Arm/Group | Flector Patch/Age 6-11 | Flector Patch/Age 12-16
Number analyzed (Participants) | 52 | 52
Participants
  No clinical improvement | 1 | 1
  Slight clinical improvement | 0 | 0
  Moderate clinical improvement | 2 | 2
  Marked clinical improvement | 2 | 9
  Normal function with no pain | 47 | 40

3. Secondary Outcome: Patient Assessment of Pain on a 6-point Scale
Description: Wong-Baker FACES Scale 6-point scale:
  No Hurt - 0; Hurts Little Bit - 1; Hurts Little More - 2; Hurts Even More - 3; Hurts Whole Lot - 4; Hurts Worst - 5.
Time Frame: Up to 2 weeks, depending upon pain resolution
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Flector Patch/Age 6-11 | Flector Patch/Age 12-16
Number analyzed (Participants) | 52 | 52
units on a scale
  Baseline | 3.37 (0.56) | 3.58 (0.64)
  Final Visit | 0.12 (0.47) | 0.27 (0.66)

4. Secondary Outcome: Plasma Concentration of Diclofenac
Time Frame: Day 2 and either Day 4, 7 or 14, depending upon pain resolution
Population: One participant missed a blood draw.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Flector Patch/Age 6-11 | Flector Patch/Age 12-16
Number analyzed (Participants) | 52 | 51
ng/mL
  24-hour | 1.83 (2.10) | 1.46 (1.88)
  Final Visit | 2.49 (3.01) | 1.11 (1.09)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 2 years and 5 months.
Arm/Group | Flector Patch/Age 6-11 | Flector Patch/Age 12-16
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/52
Other Adverse Events (participants affected / at risk) | 4/52 | 10/52
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flector Patch/Age 6-11 (N=52) | Flector Patch/Age 12-16 (N=52)
Headache (Nervous system disorders) | 4 (5) | 5 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other